CLINICAL TRIAL: NCT06428825
Title: Study in Participants With Mild to Moderate Arterial Hypertension to Investigate Safety and Tolerability of BAY3283142 in a Randomized, Single-blind, Placebo-controlled, Multi-center, Group Comparison Design
Brief Title: A Study to Learn About the Safety of BAY3283142 in People With Mild to Moderate High Blood Pressure
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Bayer (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 22723; 2024-512060-58-00 (Other: CTIS (EU))
Record Dates: First submitted 2024-05-21; First posted 2024-05-24 (Actual); Last update posted 2025-12-08 (Actual); Status verified 2025-12

CONDITIONS: Chronic Kidney Disease; Arterial Hypertension
MeSH Terms: conditions — Renal Insufficiency, Chronic; Hypertension

STUDY DESIGN:
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Treatment scheme 1 (Experimental): The Participants will receive either BAY3283142 or placebo once a day. The treatment scheme consists of 3 dose steps. Treatment will start with the low dose for 7 days , followed for 14 days at the middle dose and 14 days on the high dose.
  Interventions: Drug: BAY3283142; Drug: Placebo to BAY3283142
- Treatment scheme 2 (Experimental): Participants will receive either BAY3283142 or placebo once a day. The treatment scheme consists of 3 dose steps. Treatment will start with the low dose for 7 days , followed for 14 days at the middle dose and 7 days on the very high dose.
  Interventions: Drug: BAY3283142; Drug: Placebo to BAY3283142
- Treatment scheme 3 (Experimental): Participants will receive either BAY3283142 or placebo twice a day. The treatment scheme consists of 3 dose steps. Treatment will start with the low dose for 7 days , followed for 14 days at the middle dose and 7 days on the very high dose.
  Interventions: Drug: BAY3283142; Drug: Placebo to BAY3283142
- Treatment scheme 4 (Experimental): Participants will receive either BAY3283142 or placebo twice a day. The treatment scheme consists of 3 dose steps. Treatment will start with the low dose for 7 days , followed for 14 days at the middle dose and 14 days on the high dose.
  Interventions: Drug: BAY3283142; Drug: Placebo to BAY3283142

INTERVENTIONS:
Drug: BAY3283142 — oral administration
Drug: Placebo to BAY3283142 — oral administration

SUMMARY:
In this study, researchers want to learn about the safety of BAY3283142 after a single dose and multiple doses in participants with mild to moderate high blood pressure. The study treatment called BAY3283142 helps to relax blood vessels. It is currently under development for the treatment of chronic kidney disease (CKD). CKD is a condition in which the kidneys' ability to work gradually decrease over time. During this study, participants will take either different doses of the study drug BAY3283142 as tablets by mouth or a placebo. A placebo looks like the study drug but does not have any medicine in it. At the start of this study, the study doctor will check the medical history and current medications of the participants. They will also perform a complete health check on all the participants. Researchers will collect blood and urine samples from the participants at different time points to assess the safety and effects of BAY3283142. Each treatment scheme will consist of three doses that are given in a consecutive manner. For the first 7 days, participants will receive a lower dose of BAY3283142 in each treatment scheme. The middle and the higher dose of each treatment scheme will be given for 14 days and 7 days respectively. Participants will not know which treatment (placebo or BAY3283142) they will be given, but the study doctor will know which group received which treatment. A participant can be in the study for 10 weeks. This study will be conducted on men or postmenopausal women participants with mild to moderate high blood pressure who may not directly benefit from treatment with BAY3283142. However, information collected in this study will serve as a basis for the development of BAY3283142 for the treatment of people with CKD. Participants may experience pain and discomfort when blood samples are taken.

The researchers will closely monitor and manage any medical problems that the participants may have during the study.

ELIGIBILITY:
Inclusion Criteria:

* Participant must be 30 to 72 years of age inclusive, at the time of signing the informed consent.
* Participants with diagnosis of mild to moderate systemic arterial hypertension receiving stable treatment for ≥8 weeks before the screening visit with not more than 2 antihypertensive drugs
* No planned changes to antihypertensive treatment during active treatment phase of the study.
* Estimated glomerular filtration rate ≥45 mL/min/1.73 m2 (CKD-Epi formula) at screening and Study Day -2.
* Men and confirmed postmenopausal women (documented by medical report verification and defined as exhibiting spontaneous amenorrhea for at least 12 months before screening or as exhibiting spontaneous amenorrhea for at least 6 months before screening with documented serum follicle-stimulating hormone levels >40 miU/mL) or women with iatrogenic menopause due to bilateral oophorectomy

Exclusion Criteria:

* Systemic diseases: cancer (with the exception of appropriately treated basal cell carcinomas of the skin or uterine carcinoma in situ), autoimmune diseases (including also topically treated autoimmune diseases such as atopic dermatitis)
* Any surgical or medical condition which significantly alters the absorption, distribution, metabolism or excretion of study drugs, including, but not limited to: history of major gastrointestinal tract surgery, cholecystectomy, inflammatory bowel disease, chronic diarrhea, currently active gastritis, and pancreatitis
* Long-acting or short-acting nitrates or NO donors for any route including isosorbide dinitrate, isosorbide-5-mononitrate, pentaerythritol tetranitrate, nicorandil, nitrotriglyceride, molsidomin starting 7 days (or at least 5 half-lives of the active substance whichever is longer) before first study intervention until Follow-up.
* PDE inhibitors starting 7 days (or at least 5 half-lives of the active substance whichever is longer) before first study intervention until Follow-up.
* sGC stimulators or activators starting 7 days (or at least 5 half-lives of the active substance whichever is longer) before first study intervention until Follow-up.

Ages: 30 Years to 72 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 75 (Actual)
Dates: Start 2024-08-07 (Actual); Primary Completion 2025-11-21 (Actual); Study Completion 2025-11-21 (Actual)

PRIMARY OUTCOMES:
Number of participants with treatment-emergent adverse events per treatment arm (pooled placebo analysis) | up to 7 days after last intake of study intervention

CONTACTS AND LOCATIONS:
Locations (2):
- Germany (2):
  - Clinical Research Services | Clinical Research Services Mannheim - Phase one unit, Mannheim, Baden-Wurttemberg
  - CRS Clinical Research Services Berlin GmbH, Berlin, State of Berlin

IPD SHARING:
Plan to Share IPD: No
Availability of this study's data will later be determined according to Bayer's commitment to the EFPIA/PhRMA "Principles for responsible clinical trial data sharing". This pertains to scope, timepoint and process of data access. As such, Bayer commits to sharing upon request from qualified researchers patient-level clinical trial data, study-level clinical trial data, and protocols from clinical trials in patients for medicines and indications approved in the US and EU as necessary for conducting legitimate research. This applies to data on new medicines and indications that have been approved by the EU and US regulatory agencies on or after January 01, 2014. Interested researchers can use www.vivli.org to request access to anonymized patient-level data and supporting documents from clinical studies to conduct research. Information on the Bayer criteria for listing studies and other relevant information is provided in the member section of the portal.